CLINICAL TRIAL: NCT05312008
Title: Does Oxytocin Alter Tolerance to Alcohol or Motivation for Alcohol in Heavy Drinking Human Subjects: Testing a Novel Anti-Addiction Mechanism
Brief Title: Does Oxytocin Alter Tolerance to or Motivation for Alcohol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to complications delaying the availability of the intranasal oxytocin and IV alcohol solutions needed for this project, we were unable to complete subjects in the self-administration arm of this study.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Martin Plawecki, Associate Professor of Psychiatry, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 10002
Record Dates: First submitted 2022-02-26; First posted 2022-04-05 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol use disorder; Oxytocin, intranasal; Alcohol tolerance; Alcohol intake; Alcohol treatment; Alcohol, intravenous
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: 2 Arms; both 2 session crossover design
Who Masked: Participant, Investigator
Masking Description: The pharmacy will prepare the intranasal spray (both oxytocin and placebo) and deliver it in coded syringes to the lab. Investigators, laboratory staff and subjects will be unaware of the identity of the spray on session days. The pharmacy will provide the unmasking information after all sessions are completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clamp (Experimental): Repeated subjective and cognitive tests during a 4 hour session that includes a baseline period, an oxytocin or placebo delivery, absorption and testing period, and a 2 hour alcohol clamp. Oxytocin or placebo were delivered intranasally in two sessions, scheduled 3-4 weeks apart, double blind.
  Interventions: Drug: Intranasal oxytocin; Drug: Intranasal placebo
- Progressive work for alcohol (Experimental): Progressive work alcohol exposure, 2 sessions (intranasal oxytocin or placebo), double blind.
  Note this Arm was not completed (see Overall Status for explanation of study termination)
  Interventions: Drug: Intranasal oxytocin; Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intranasal oxytocin — Initial dose 40 IU in 1 ml; 2 booster doses of 24 IU in 0.6 mls each, spaced about 1 hour apart
Drug: Intranasal placebo — Initial volume 1 ml; 2 booster volumes of 0.6 mls each, spaced about 1 hour apart

SUMMARY:
This pilot study is intended to demonstrate feasibility and acquire preliminary data. If successful, this data could support a future project studying the effect of oxytocin on tolerance and alcohol seeking in humans.

DETAILED DESCRIPTION:
This pilot study is designed to demonstrate feasibility and provide preliminary data supporting use of intranasal oxytocin in treatment of alcohol use disorders. Specifically, experiments are planned to test the ability of oxytocin to reverse tolerance and alcohol seeking in humans by employing state-of-the-art computer-assisted intravenous alcohol administration. Two separate experiments will be run. In the first, tolerance will be assessed using sensitive tests of subjective response and cognitive function during an intravenous infusion that maintains a steady breath and therefore brain exposure to alcohol. In the second, an intravenous alcohol self-administration paradigm that requires increasing effort for each additional infusion will be used to assess change in motivation for alcohol. Demonstrating that oxytocin (compared to placebo) worsens test performances in alcohol-dependent individuals and/or reduces the compulsive drive to self-administer alcohol would be strong evidence for its potential to treat alcohol use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Heavy alcohol drinkers.
* Able to understand/complete questionnaires and procedures in English.
* Have venous access sufficient to allow blood sampling.

Exclusion Criteria:

* Latex allergy.
* Nasal condition that compromises delivery and/or absorption of intra-nasal oxytocin
* Pregnant or breast-feeding women.
* Desire to be treated for any substance use disorder or court ordered to not drink alcohol
* Medical disorders or other conditions such as alcohol withdrawal seizures or delirium tremens that may influence study outcome or participant safety.
* Positive urine drug screen for amphetamines/ methamphetamines, barbiturates, benzodiazepines, cocaine, opiates, or phencyclidine if determined by the PI to adversely affect participant safety or data integrity.
* Medications (past 30 days) that could influence participant safety or data integrity (e.g. antidepressants, antipsychotics, benzodiazepines, etc.) as determined by the PI.
* DSM 5 Disorders (other than alcohol) or current/history of neurological disease of cerebral origin, or head injury with > 20 min loss of consciousness, if determined by the PI to affect participant safety or data integrity.
* Positive breath alcohol reading at beginning of the experimental session.
* Actively suicidal (for example, any current suicidal intent, including a plan) or are at serious suicidal risk, by clinical judgment of the PI.
* Any condition for which the PI and investigative team determine it is unsafe or not prudent to enroll a participant.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-01-16 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Plawecki, MD, PhD, Principal Investigator — Psychiatry, Indiana University School of Medicine
Locations (1):
- University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The final raw dataset will be available to other researchers when we have collected all subjects, completed our own planned analyses, and, if warranted, sought and obtained funding based on the outcome of this pilot study.
Supporting Information: Study Protocol, ICF
Time Frame: The dataset will be available indefinitely
Access Criteria: On request to the PI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were contacted from our lab's recruiting database. Recruiting was active between January and May, 2022, and between October and November, 2023.
Pre-assignment Details: Due to complications delaying the availability of the intranasal oxytocin and IV alcohol solutions needed for this project, we were unable to complete subjects in the self-administration arm of this study
Groups:
- Oxytocin First, Then Placebo (Clamp); Placebo First, Then Oxytocin (Clamp): Clamped alcohol exposure, repeated tests of subjective and cognitive effects of alcohol, 2 sessions (intranasal oxytocin or placebo), double blind
  Intranasal oxytocin: Initial dose 40 IU in 1 ml; 2 booster doses of 24 IU in 0.6 mls each, spaced about 1 hour apart
  Intranasal placebo: Initial volume 1 ml; 2 booster volumes of 0.6 mls each, spaced about 1 hour apart
- Oxytocin First, Then Placebo (Progressive Work); Placebo First, Then Oxytocin (Progressive Work): Session in which participants could self-administer brief infusions of alcohol solutions. Opportunities for infusions could be earned by completing repetitions of a constant-attention button pressing task; the number of completions required increased over time (a progressive work schedule).
  Note no participants were enrolled in this Arm (see project termination for explanation).
Period: Overall Study
Arm/Group | Oxytocin First, Then Placebo (Clamp) | Placebo First, Then Oxytocin (Clamp) | Oxytocin First, Then Placebo (Progressive Work) | Placebo First, Then Oxytocin (Progressive Work)
Started | 3 | 3 | 0 | 0
Completed | 3 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants in this study
Groups:
- All Participants: Demographic information is provided for all 6 participants combined. All 6 subjects participated in the clamp arm. The self-administration arm was not completed (see Overall Status). 3 participants had the Oxytocin session first, then Placebo; the other 3 had the reverse order (Placebo then Oxytocin).
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Subjective Effect of Alcohol - Craving
Description: Participants rated their subjective feeling of craving on a scale of 0-100. Tolerance to alcohol is assessed by subtracting subjective ratings at the beginning of the 2 hour alcohol infusion from ratings at the end; a negative value indicates tolerance. Possible scores ranged from -100 to 100; negative scores indicate the development of tolerance. Values reported here compare tolerance developed during the oxytocin session to tolerance developed during the placebo session.
Time Frame: 2 single day laboratory sessions, one with intranasal oxytocin, one with intranasal placebo, scheduled 3-4 weeks apart, order counter-balanced.
Population: All participants who completed both the oxytocin and placebo sessions were included.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Oxytocin Session (Clamp): Measurements acquired during the Oxytocin Session
- Placebo Session (Clamp): Measurements acquired during the placebo session
Arm/Group | Oxytocin Session (Clamp) | Placebo Session (Clamp)
Number analyzed (Participants) | 6 | 6
units on a scale | 1.6 (11.4) | 10.5 (10.3)
Statistical Analysis 1: Comparison: Oxytocin Session (Clamp) vs Placebo Session (Clamp); Test type: Superiority; p < 0.6, t-test, 2 sided; paired

2. Primary Outcome: Subjective Effects of Alcohol - Intoxication
Description: Participants rated their subjective feeling of intoxication on a scale of 0-100. Tolerance to alcohol is assessed by subtracting subjective ratings at the beginning of the 2 hour alcohol infusion from ratings at the end. Using this calculation, theoretical scores in this dataset could range from -100-100; negative scores indicate the development of tolerance. Values reported here compare tolerance developed during the oxytocin session to tolerance developed during the placebo session.
Time Frame: as for outcome 1
Population: All participants who completed both the Oxytocin and Placebo sessions are included in the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oxytocin Session (Clamp) | Placebo Session (Clamp)
Number analyzed (Participants) | 6 | 6
units on a scale | 1.0 (7.8) | 7.8 (13.2)
Statistical Analysis 1: Comparison: Oxytocin Session (Clamp) vs Placebo Session (Clamp); Test type: Superiority; p < 0.6, t-test, 2 sided; Paired

3. Primary Outcome: Stop Signal Response Task
Description: The Stop Signal task asks participants to respond as quickly as they can to one stimulus (the "Go" signal) but withhold this response when a second, much rarer stimulus appears (the "Stop" signal). Performance reported here uses the variable ssRT Med, which is an estimate of the time (in ms) needed to stop and withdraw the response; alcohol is known to increase ssRT Med. To assess tolerance, the value of ssRT Med measured at the beginning of the 2 hour alcohol clamp was subtracted from the value measured at the end. The theoretical range of possible scores on this measure range from about -100 to 200; negative scores indicate the development of tolerance. Values reported here compare tolerance developed during the oxytocin session to tolerance developed during the placebo session.
Time Frame: as for outcome 1
Population: All participants who completed both the Oxytocin and Placebo sessions are included in the analysis.
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Oxytocin Session (Clamp) | Placebo Session (Clamp)
Number analyzed (Participants) | 6 | 6
milliseconds | -1.8 (18) | -1.1 (8)
Statistical Analysis 1: Comparison: Oxytocin Session (Clamp) vs Placebo Session (Clamp); Test type: Superiority; p < 1, t-test, 2 sided; Paired

4. Primary Outcome: Stroop Test
Description: The Stroop Interference task asks participants to respond to one aspect of a stimulus (in this case, the color of the text in which a word is printed) under conditions in which the word meaning either enhances or interferes with the task (for example, the word Green in a Green font speeds performance, while the word Green in a Yellow font slows performance). Tolerance to alcohol was assessed by subtracting response latency (ms) on correct trials at the beginning of the 2 hour alcohol infusion from latency on correct trials at the end. Theoretical scores ranged from about -200 to 250; negative scores indicate the development of tolerance. Values reported here compare tolerance developed during the oxytocin session to tolerance developed during the placebo session.
Time Frame: as for outcome 1
Population: All participants who completed both the Oxytocin and Placebo sessions are included in the analysis.
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Oxytocin Session (Clamp) | Placebo Session (Clamp)
Number analyzed (Participants) | 6 | 6
milliseconds | -1.56 (13.3) | -29.82 (13.1)
Statistical Analysis 1: Comparison: Oxytocin Session (Clamp) vs Placebo Session (Clamp); Test type: Superiority; p < 0.04, t-test, 2 sided; Paired

5. Primary Outcome: Alcohol Purchase Task (Variable OMax)
Description: The Alcohol Purchase task (APT) tests the value participants place on alcohol at specific times and conditions of the experimental session. To complete the APT, participants fill out a table reporting how many drinks (allowed range 0-50) they would purchase during an evening out, for a cost ranging from $0 to $30/drink. From this, a value for # of drinks * cost of drink is calculated; OMax is the highest amount in dollars that a participant would spend (possible range = $0 to $1,500). Tolerance to the effect of alcohol is calculated as OMax (end of infusion) - OMax (beginning of infusion), possible values range from -$1,500 to $1,500. Negative scores indicate the development of tolerance. Values reported here compare tolerance developed during the oxytocin session to tolerance developed during the placebo session.
Time Frame: 2 single day laboratory sessions, one with intranasal oxytocin, one with intranasal placebo
Population: All participants who completed both the Oxytocin and Placebo sessions are included in the analysis.
Measure: Mean (Standard Error); unit: dollars
Arm/Group | Oxytocin Session (Clamp) | Placebo Session (Clamp)
Number analyzed (Participants) | 6 | 6
dollars | -1.0 (2.1) | -3.2 (2.2)
Statistical Analysis 1: Comparison: Oxytocin Session (Clamp) vs Placebo Session (Clamp); Test type: Superiority; p < 0.5, t-test, 2 sided; Paired

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during 3 time periods: Oxytocin session day (~12 hours from arrival at to dismissal from Clinical Research Center) Between session day interval (21-28 days) Placebo session day (~12 hours from arrival at to dismissal from Clinical Research Center)
Description: Adverse event data were collected during the sessions by tracking expected oxytocin side-effects at each testing block. Specific symptoms monitored included dizziness, dry mouth, runny nose, stomach pain, nausea, headache, or any other unusual feeling.
  Adverse events were also collected unsystematically by asking the subject to report on their wellbeing and any unusual symptoms at study day intake, during the session, and during the post-session recovery period (3-6 hours).
Groups:
- Oxytocin Session: Measurements acquired during the Oxytocin Session
- Placebo: Measurements acquired during the placebo session
- Between Session Interval: Events occurring between the first and second session day
Arm/Group | Oxytocin Session | Placebo | Between Session Interval
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 4/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin Session (N=6) | Placebo (N=6) | Between Session Interval (N=6)
Nausea (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 4 (4) | 0 (0)
Infected Toe (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Participant reported an active toe infection at session 2 that began sometime after session 1; was treated by physician. PI determined the infection was not related to study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT05312008/Prot_SAP_000.pdf